CLINICAL TRIAL: NCT02979613
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of Switching From Tenofovir Disoproxil Fumarate (TDF) 300 mg QD to Tenofovir Alafenamide (TAF) 25 mg QD in Subjects With Chronic Hepatitis B Who Are Virologically Suppressed
Brief Title: Study to Evaluate Efficacy and Safety of Switching From TDF to TAF in Adults With Chronic Hepatitis B Who Are Virologically Suppressed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-320-4018; 2016-003632-20 (EudraCT Number)
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-08

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAF 25 mg (Experimental): Double-blind (DB) phase: TAF 25 mg + TDF placebo for up to 53 weeks. Open-label extension (OLE) phase: TAF 25 mg for up to 52 weeks.
  Interventions: Drug: TAF; Drug: TDF Placebo
- TDF 300 mg (Active Comparator): DB phase: TDF 300 mg + TAF placebo for up to 50 weeks. OLE phase: TAF 25 mg for up to 52 weeks.
  Interventions: Drug: TAF; Drug: TDF; Drug: TAF Placebo

INTERVENTIONS:
Drug: TAF — 25 mg tablet administered orally once daily
  Other Names: Vemlidy®; GS-7340
Drug: TDF — 300 mg tablet administered orally once daily
  Other Names: Viread®
  Arms: TDF 300 mg
Drug: TAF Placebo — Tablet administered orally once daily
  Arms: TDF 300 mg
Drug: TDF Placebo — Tablet administered orally once daily
  Arms: TAF 25 mg

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of switching to tenofovir alafenamide (TAF) versus continuing tenofovir disoproxil fumarate (TDF) in virologically suppressed adults with chronic hepatitis B virus (HBV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent form; consent must be obtained prior to initiation of study procedures
* Adult male and non-pregnant, non-lactating females
* Documented evidence of chronic hepatitis B virus (HBV) infection previously
* Maintained on tenofovir disoproxil fumarate (TDF) 300 mg once daily for at least 48 weeks, and as monotherapy for chronic hepatitis B for at least 24 weeks with viral suppression (HBV DNA < lower limit of quantitation) for a minimum of 12 weeks prior to screening
* Adequate renal function
* Normal Electrocardiogram

Key Exclusion Criteria:

* Pregnant women or women who are breastfeeding
* Males and females of reproductive potential who are unwilling to use an "effective", protocol-specified method(s) of contraception during the study.
* Co-infection with hepatitis C virus (HCV), hepatitis D virus (HDV), or human immunodeficiency virus (HIV)
* Evidence of hepatocellular carcinoma
* Current evidence of, or recent (≤ 5 year) history of clinical hepatic decompensation
* Abnormal hematological and biochemical parameters, including:

  * Hemoglobin < 10 g/dL
  * Absolute neutrophil count < 750/mm^3
  * Platelets ≤ 50,000/mm^3
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 × upper limit of the normal (ULN)
  * Albumin < 3.0 mg/ dL
  * International normalized ratio (INR) > 1.5 × ULN (unless stable on anticoagulant regimen)
  * Total bilirubin > 2.5 × ULN
* Received solid organ or bone marrow transplant
* Malignancy within 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (eg, basal cell skin cancer). Individuals under evaluation for possible malignancy are not eligible.
* Currently receiving therapy with immunomodulators (eg, corticosteroids), nephrotoxic agents, or agents capable of modifying renal excretion
* Individuals receiving ongoing therapy with drugs not to be used with TAF or TDF or individuals with a known hypersensitivity to study drugs, metabolites, or formulation excipients
* Current alcohol or substance abuse judged by the investigator to potentially interfere with compliance
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the individual unsuitable for the study or unable to comply with dosing requirements.
* Use of investigational agents within 3 months of screening, unless allowed by the sponsor

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (29):
- United States (14):
  - Los Angeles, California
  - Palo Alto, California
  - Pasadena, California
  - San Diego, California
  - San Francisco, California
  - San Jose, California
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Novi, Michigan
  - Flushing, New York
  - New York, New York
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Sugar Land, Texas
- Canada (3):
  - Edmonton
  - Toronto
  - Vancouver
- Hong Kong (2):
  - Hong Kong
  - Kowloon
- Milan, Italy
- South Korea (3):
  - Goyang, Gyeonggi-d
  - Daegu
  - Seoul
- Spain (2):
  - Barcelona
  - Majadahonda
- Taiwan (3):
  - Chiayi City
  - Kaohsiung City
  - Taipei
- London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Lampertico P, Buti M, Fung S, Ahn SH, Chuang WL, Tak WY, Ramji A, Chen CY, Tam E, Bae H, Ma X, Flaherty JF, Gaggar A, Lau A, Liu Y, Wu G, Suri V, Tan SK, Subramanian GM, Trinh H, Yoon SK, Agarwal K, Lim YS, Chan HLY. Switching from tenofovir disoproxil fumarate to tenofovir alafenamide in virologically suppressed patients with chronic hepatitis B: a randomised, double-blind, phase 3, multicentre non-inferiority study. Lancet Gastroenterol Hepatol. 2020 May;5(5):441-453. doi: 10.1016/S2468-1253(19)30421-2. Epub 2020 Feb 20. PMID 32087795

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and Asia. The first participant was screened on 29 December 2016. The last study visit occurred on 30 January 2020.
Pre-assignment Details: 541 participants were screened.
Groups:
- TAF 25 mg: Participants who were virologically suppressed and taking tenofovir disoproxil fumarate (TDF) 300 mg tablet orally once daily received tenofovir alafenamide (TAF) 25 mg tablet orally once daily, and placebo to match TDF once daily for up to 53 weeks in the double-blind (DB) phase. Participants who completed DB treatment and were willing to enter in the open-label extension (OLE) phase, received TAF 25 mg tablet orally once daily for up to 52 weeks.
- TDF 300 mg: Participants who were virologically suppressed and taking TDF 300 mg tablet orally once daily received TDF 300 mg tablet orally once daily, and placebo to match TAF once daily for up to 50 weeks in the DB phase. Participants who completed DB treatment and were willing to enter in the OLE phase, received TAF 25 mg tablet orally once daily for up to 52 weeks.
Period: Double-Blind Phase
Arm/Group | TAF 25 mg | TDF 300 mg
Started | 245 | 245
Completed | 235 | 237
Not Completed | 10 | 8
Not completed — Withdrew Consent | 2 | 4
Not completed — Pregnancy | 2 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Randomized but Never Treated | 2 | 0
Period: Open-Label Extension (OLE) Phase
Arm/Group | TAF 25 mg | TDF 300 mg
Started | 235 | 237
Completed | 232 | 231
Not Completed | 3 | 6
Not completed — Withdrew Consent | 2 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1
Not completed — Investigator's Discretion | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all randomized participants who received at least 1 dose of study drug.
Groups:
- TAF 25 mg: Participants who were virologically suppressed and taking TDF 300 mg tablet orally once daily received TAF 25 mg tablet orally once daily, and placebo to match TDF once daily for up to 53 weeks in the DB phase. Participants who completed DB treatment and were willing to enter in the OLE phase, received TAF 25 mg tablet orally once daily for up to 52 weeks.
- Total: Total of all reporting groups
Arm/Group | TAF 25 mg | TDF 300 mg | Total
Number analyzed (Participants) | 243 | 245 | 488
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (10.5) | 51 (10.8) | 51 (10.7)
Age, Customized [Count of Participants; unit: Participants]
  < 50 Years | 107 | 109 | 216
  ≥ 50 Years | 136 | 136 | 272
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 79 | 143
  Male | 179 | 166 | 345
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 240 | 245 | 485
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 195 | 205 | 400
  Race: Black or African American | 9 | 8 | 17
  Race: Native Hawaiian or Pacific Islander | 0 | 1 | 1
  Race: White | 38 | 31 | 69
  Race: Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 42 | 47 | 89
  South Korea | 61 | 77 | 138
  Hong Kong | 15 | 13 | 28
  United States | 63 | 64 | 127
  Taiwan | 28 | 13 | 41
  Italy | 9 | 12 | 21
  United Kingdom | 6 | 7 | 13
  Spain | 19 | 12 | 31
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: U/L] | 28 (15.6) | 26 (12.0) | 27 (13.9)
ALT Level Based on Central Lab Normal Range [Count of Participants; unit: Participants] — Central laboratory upper limit of normal (ULN) for ALT were as follows: ≤ 43 U/L for males aged 18 to < 69 years and ≤ 35 U/L for males aged ≥ 69 years; ≤ 34 U/L for females aged 18 to < 69 years and ≤ 32 U/L for females aged ≥ 69 years.
  Participants
    ≤ ULN | 211 | 226 | 437
    > ULN to 5xULN | 32 | 19 | 51
    > 5xULN | 0 | 0 | 0
ALT Level Based on 2018 American Association for the Study of Liver Diseases (AASLD) Normal Range [Count of Participants; unit: Participants] — The ULN for ALT using the 2018 AASLD normal range was 25 U/L for females and 35 U/L for males.
  Participants
    ≤ ULN | 191 | 192 | 383
    > ULN to 5xULN | 52 | 53 | 105
    > 5xULN | 0 | 0 | 0
Hepatitis B virus (HBV) DNA Category [Count of Participants; unit: Participants]
  < 20 IU/mL | 238 | 242 | 480
  20 to < 69 IU/mL | 2 | 3 | 5
  ≥ 69 IU/mL | 3 | 0 | 3
Hepatitis B e Antigen/Antibody (HBeAg/HBeAb) Status [Count of Participants; unit: Participants] — HBeAb status was imputed as negative if missing.
  Participants
    Positive/Negative | 78 | 78 | 156
    Positive/Positive | 0 | 1 | 1
    Negative/Negative | 17 | 28 | 45
    Negative/Positive | 148 | 138 | 286
FibroTest® Score [Mean (Standard Deviation); unit: scores on a scale] — The FibroTest® score is used to assess liver fibrosis. Scores range from 0.00 to 1.00, with higher scores indicating a greater degree of fibrosis. Population: Participants in Safety Analysis Set with available data were analyzed.
  scores on a scale
    number analyzed (Participants) | 241 | 245 | 486
    (all) | 0.42 (0.234) | 0.41 (0.211) | 0.42 (0.223)
Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFR-CG) [Mean (Standard Deviation); unit: mL/min] | 95.0 (25.58) | 93.8 (25.16) | 94.4 (25.35)
Hip Bone Mineral Density (BMD) Status [Count of Participants; unit: Participants] — Population: Hip Dual-Energy X-Ray Absorptiometry (DXA) Analysis Set included all participants who were randomized into the study, received at least 1 dose of study drug, and had nonmissing baseline hip BMD values.
  Participants
    number analyzed (Participants) | 241 | 244 | 485
    Normal (T-score ≥ -1.0) | 143 | 124 | 267
    Osteopenia (-2.5 ≤ T-score < -1.0) | 89 | 116 | 205
    Osteoporosis (T-score < -2.5) | 9 | 4 | 13
Spine BMD Status [Count of Participants; unit: Participants] — Spine DXA Analysis Set included all participants who were randomized into the study, received at least 1 dose of study drug, and had nonmissing baseline spine BMD values.
  Participants
    Normal (T-score ≥ -1.0) | 125 | 120 | 245
    Osteopenia (-2.5 ≤ T-score < -1.0) | 90 | 97 | 187
    Osteoporosis (T-score < -2.5) | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis B Virus (HBV) DNA Levels ≥ 20 IU/mL at Week 48, as Determined by the Modified United States Food and Drug Administration (US FDA)-Defined Snapshot Algorithm
Description: The percentage of participants with HBV DNA ≥ 20 IU/mL at Week 48 was analyzed using the modified US FDA-defined snapshot algorithm, which included participants who:
  1. Had the last available on-treatment HBV DNA ≥ 20 IU/mL in the Week 48 analysis window (from Day 295 to Day 378, inclusive), or
  2. Did not have on-treatment HBV DNA data available in the Week 48 analysis window and
     * Discontinued study drug prior to or in the Week 48 analysis window due to lack of efficacy, or
     * Discontinued study drug prior to or in the Week 48 analysis window due to reason other than lack of efficacy and had the last available on-treatment HBV DNA ≥ 20 IU/mL
Time Frame: Week 48
Population: The Full Analysis Set included all participants who were randomized into the study and received at least 1 dose of study drug. Participants were analyzed according to the treatment to which they were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 243 | 245
percentage of participants | 0.4 | 0.4
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; The null hypothesis was that the TAF group is at least 4% worse than the TDF group with respect to the percentage of participants with HBV DNA ≥ 20 IU/mL at Week 48. The alternative hypothesis was that the TAF group is less than 4% worse than the TDF group with respect to the percentage of participants with HBV DNA ≥ 20 IU/mL at Week 48; Test type: Non-Inferiority — Non-inferiority was assessed using a 95% confidence interval (CI) approach, with a non-inferiority margin of 4%; Difference in the Percentages = 0.0, 95% CI 2-sided [-1.9 to 2.0] — Difference in the percentages of participants between treatment groups and its 95% CI were calculated based on the stratum-adjusted Mantel-Haenszel (MH) percentage, adjusted by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata

2. Secondary Outcome: Percentage of Participants With HBV DNA Levels ≥ 20 IU/mL at Week 96, as Determined by the Modified US FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HBV DNA ≥ 20 IU/mL at Week 96 was analyzed using the modified US FDA-defined snapshot algorithm, which included participants who:
  1. Had the last available on-treatment HBV DNA ≥ 20 IU/mL in the Week 96 analysis window (from Day 589 to Day 840, inclusive), or
  2. Did not have on-treatment HBV DNA data available in the Week 96 analysis window and
     * Discontinued study drug prior to or in the Week 96 analysis window due to lack of efficacy, or
     * Discontinued study drug prior to or in the Week 96 analysis window due to reason other than lack of efficacy and had the last available on-treatment HBV DNA ≥ 20 IU/mL
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed. Participants were analyzed according to the treatment to which they were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 243 | 245
percentage of participants | 0.4 | 0.4
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Non-Inferiority — Non-inferiority was assessed using a 95% confidence interval (CI) approach, with a non-inferiority margin of 4%; Difference in the Percentages = 0.0, 95% CI 2-sided [-1.9 to 1.9] — Difference in the percentage of participants between treatment groups and its 95% CI were calculated based on the stratum-adjusted MH percentage, adjusted by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata
Statistical Analysis 2: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Superiority; p = 0.9953, Cochran-Mantel-Haenszel — P-value for the superiority tests compared the percentage of each HBV DNA outcome was from CMH tests stratified by baseline age groups and baseline HBeAg status strata

3. Secondary Outcome: Percentage of Participants With HBV DNA Levels < 20 IU/mL at Week 48
Description: The percentage of participants with HBV DNA < 20 IU/mL at Week 48 was analyzed, which included participants who have the last available on-treatment HBV DNA, 20 IU/mL in the Week 48 analysis window. Missing=Failure (M = F) approach was used for analysis.
Time Frame: Weeks 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 243 | 245
percentage of participants | 96.3 | 96.3
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Non-Inferiority — Non-inferiority was assessed using a 95% CI approach, with a non-inferiority margin of 4%; Difference in the Percentages = -0.0, 95% CI 2-sided [-3.7 to 3.7] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Superiority; p = 0.98, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 2]

4. Secondary Outcome: Percentage of Participants With HBV DNA Levels < 20 IU/mL (Target Detected/Not Detected) at Week 48
Description: The percentage of participants with HBV DNA < 20 IU/mL at Week 48 was analyzed, which included participants who have the last available on-treatment HBV DNA, 20 IU/mL in the Week 48 analysis window. The method of determining percentage of participants with HBV DNA levels <20 IU/mL (target detected/not detected i.e., lower limit of detection) at Week 48, was handled by M = F, and Missing=Excluded (M = E) approaches.
Time Frame: Week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 243 | 245
percentage of participants
  M = F Approach: < 20 IU/mL Target Not Detected | 63.4 | 62.0
  M = F Approach: < 20 IU/mL Target Detected | 32.9 | 34.3
  M = E Approach: < 20 IU/mL Target Not Detected | 65.5 | 64.1
  M = E Approach: < 20 IU/mL Target Detected | 34.0 | 35.4

5. Secondary Outcome: Percentage of Participants With HBV DNA Levels < 20 IU/mL at Week 96
Description: The percentage of participants with HBV DNA < 20 IU/mL at Week 96 was analyzed, which included participants who have the last available on-treatment HBV DNA, 20 IU/mL in the Week 96 analysis window. M = F approach was used for analysis.
Time Frame: Week 96
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 243 | 245
percentage of participants | 94.7 | 93.9
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Non-Inferiority — Non-inferiority was assessed using a 95% confidence interval (CI) approach, with a non-inferiority margin of 4%; Difference in the Percentages = 0.9, 95.0% CI 2-sided [-3.5 to 5.2] — Difference in the percentages of participants between treatment groups and its 95% CI were calculated based on the stratum-adjusted MH percentage, adjusted by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata
Statistical Analysis 2: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Superiority; p = 0.6863, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 2]

6. Secondary Outcome: Percentage of Participants With HBV DNA Levels < 20 IU/mL (Target Detected/Not Detected) at Week 96
Description: The percentage of participants with HBV DNA < 20 IU/mL at Week 96 was analyzed, which included participants who have the last available on-treatment HBV DNA, 20 IU/mL in the Week 96 analysis window. The method of determining percentage of participants with HBV DNA levels <20 IU/mL (target detected/not detected i.e., lower limit of detection) at Week 96, was handled by Missing=Failure (M = F), and Missing=Excluded (M = E) approaches.
Time Frame: Week 96
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 243 | 245
percentage of participants
  M = F Approach: < 20 IU/mL Target Not Detected | 65.8 | 66.1
  M = F Approach: < 20 IU/mL Target Detected | 28.8 | 27.8
  M = E Approach: < 20 IU/mL Target Not Detected | 69.3 | 70.1
  M = E Approach: < 20 IU/mL Target Detected | 30.3 | 29.4

7. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Loss at Week 48
Description: HBeAg loss was defined as HBeAg changing from positive at baseline to negative at a postbaseline visit with baseline HBeAb negative or missing. The M = F approach was used for this analysis.
Time Frame: Week 48
Population: The Serologically Evaluable Full Analysis Set for HBeAg loss and seroconversion included all participants who were randomized and received at least 1 dose of study drug and were HBeAg-positive and HBeAb-negative or had a missing value at baseline. Participants were analyzed according to the treatment to which they were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 78 | 78
percentage of participants | 7.7 | 6.4
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Superiority; p = 0.7258, Cochran-Mantel-Haenszel — P-value was from the CMH test, stratified by baseline age groups (< 50, ≥ 50 years); Difference in the Percentages = 1.4, 95% CI 2-sided [-7.2 to 10.1] — Difference in the percentage of participants between the treatment groups and its 95% CI were calculated based on the stratum-adjusted MH percentage, adjusted by baseline age groups

8. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion at Week 48
Description: HBeAg seroconversion was defined as HBeAg loss and HBeAb changing from negative/missing at baseline to positive at a postbaseline visit. The M = F approach was used for this analysis.
Time Frame: Week 48
Population: Participants in the Serologically Evaluable Full Analysis Set for HBeAg loss and seroconversion were analyzed. Participants were analyzed according to the treatment to which they were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 78 | 78
percentage of participants | 2.6 | 0.0
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Superiority; p = 0.1348, Cochran-Mantel-Haenszel — P-value was from the CMH test, stratified by baseline age groups (< 50, ≥ 50 years); Difference in the Percentages = 2.7, 95% CI 2-sided [-2.3 to 7.7] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Percentage of Participants With HBeAg Loss at Week 96
Description: as for outcome 7
Time Frame: Week 96
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 78 | 78
percentage of participants | 17.9 | 9.0
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Superiority; p = 0.1005, Cochran-Mantel-Haenszel — P-value was from CMH tests stratified by baseline age groups (< 50, ≥ 50 years); Difference in the Percentages = 9.0, 95% CI 2-sided [-2.0 to 20.1] — Difference in the percentages of participants between treatment groups and its 95% CI were calculated based on the stratum-adjusted MH percentage, adjusted by baseline age groups

10. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion at Week 96
Description: as for outcome 8
Time Frame: Week 96
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 78 | 78
percentage of participants | 5.1 | 2.6
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Superiority; p = 0.4154, Cochran-Mantel-Haenszel — P-value was from CMH tests stratified by baseline age groups (< 50, ≥ 50 years); Difference in the Percentages = 2.5, 95% CI 2-sided [-4.5 to 9.5] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Loss at Week 48
Description: HBsAg loss was defined as HBsAg changing from positive at baseline to negative at a postbaseline visit with baseline HBsAb negative or missing. The M = F approach was used for this analysis.
Time Frame: Week 48
Population: The Serologically Evaluable Full Analysis Set for HBsAg loss and seroconversion included all participants who were randomized and received at least 1 dose of study drug and were HBsAg-positive and HBsAb-negative or had a missing value at baseline. Participants were analyzed according to the treatment to which they were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 243 | 245
percentage of participants | 0.0 | 2.0
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Superiority; p = 0.0281, Cochran-Mantel-Haenszel — P-value was from the CMH test, stratified by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata; Difference in the Percentages = -2.0, 95% CI 2-sided [-4.4 to 0.3] — Difference in the percentage of participants between the treatment groups and its 95% CI were calculated based on the stratum-adjusted MH percentage, adjusted by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata

12. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at Week 48
Description: HBsAg seroconversion was defined as HBsAg loss and HBsAb changes from negative/missing at baseline to positive at a postbaseline visit. The M = F approach was used for this analysis.
Time Frame: Week 48
Population: Participants in the Serologically Evaluable Full Analysis Set for HBsAg loss and seroconversion were analyzed. Participants were analyzed according to the treatment to which they were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 243 | 245
percentage of participants | 0.0 | 0.0

13. Secondary Outcome: Percentage of Participants With HBsAg Loss at Week 96
Description: as for outcome 11
Time Frame: Week 96
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 243 | 245
percentage of participants | 1.6 | 2.4
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Superiority; p = 0.5373, Cochran-Mantel-Haenszel — P-value was from CMH tests stratified by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata; Difference in the Percentages = -0.8, 95% CI 2-sided [-3.7 to 2.1] — [estimate comment as in outcome 5, analysis 1]

14. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at Week 96
Description: as for outcome 12
Time Frame: Week 96
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 243 | 245
percentage of participants | 0.8 | 0.4
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Superiority; p = 0.5845, Cochran-Mantel-Haenszel — P-value was from CMH tests stratified by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata; Difference in the Percentages = 0.4, 95% CI 2-sided [-1.7 to 2.5] — [estimate comment as in outcome 5, analysis 1]

15. Secondary Outcome: Percentage of Participants With Normal Alanine Aminotransferase (ALT) at Week 48 (by Central Laboratory and the American Association for the Study of Liver Diseases [AASLD] Criteria)
Description: Central laboratory ULN for ALT were as follows: ≤ 43 U/L for males aged 18 to < 69 years and ≤ 35 U/L for males aged ≥ 69 years; ≤ 34 U/L for females aged 18 to < 69 years and ≤ 32 U/L for females aged ≥ 69 years. The ULN for ALT using the 2018 AASLD normal range was 25 U/L for females and 35 U/L for males. M = F approach was used for analysis.
Time Frame: Week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 243 | 245
percentage of participants
  Central Laboratory Criteria | 89.3 | 84.9
  AASLD Criteria | 79.0 | 75.1
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Central Laboratory Criteria; Test type: Superiority; p = 0.1405, Cochran-Mantel-Haenszel — P-value was from the CMH test, stratified by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata; Difference in the Percentages = 4.5, 95% CI 2-sided [-1.6 to 10.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: TAF 25 mg vs TDF 300 mg; AASLD Criteria; Test type: Superiority; p = 0.3133, Cochran-Mantel-Haenszel — P-value was from the CMH test, stratified by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata; Difference in the Percentages = 3.8, 95% CI 2-sided [-3.7 to 11.4] — [estimate comment as in outcome 11, analysis 1]

16. Secondary Outcome: Percentage of Participants With Normalized ALT at Week 48 (by Central Laboratory and AASLD Criteria)
Description: ALT normalization was defined as an ALT value that changed from above the normal range at baseline to within the normal range at the given postbaseline visit. Central laboratory ULN for ALT were as follows: ≤ 43 U/L for males aged 18 to < 69 years and ≤ 35 U/L for males aged ≥ 69 years; ≤ 34 U/L for females aged 18 to < 69 years and ≤ 32 U/L for females aged ≥ 69 years. The ULN for ALT using the 2018 AASLD normal range was 25 U/L for females and 35 U/L for males. M = F approach was used for analysis.
Time Frame: Week 48
Population: Participants in the Full Analysis Set with Baseline ALT > ULN were analyzed. Participants were analyzed according to the treatment to which they were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 52 | 53
percentage of participants
  Central Laboratory Criteria: number analyzed (Participants) | 32 | 19
  Central Laboratory Criteria | 50.0 | 36.8
  AASLD Criteria | 50.0 | 26.4
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Central Laboratory criteria; Test type: Superiority; p = 0.3381, Cochran-Mantel-Haenszel — P-value was from the CMH test, stratified by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata; Difference in the Percentages = 14.1, 95% CI 2-sided [-16.4 to 44.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: TAF 25 mg vs TDF 300 mg; AASLD Criteria; Test type: Superiority; p = 0.0136, Cochran-Mantel-Haenszel — P-value was from the CMH test, stratified by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata; Difference in the Percentages = 23.8, 95% CI 2-sided [5.3 to 42.3] — [estimate comment as in outcome 11, analysis 1]

17. Secondary Outcome: Percentage of Participants With Normal ALT at Week 96 (by Central Laboratory and the AASLD Criteria)
Description: as for outcome 15
Time Frame: Week 96
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 243 | 245
percentage of participants
  Central Laboratory Criteria | 88.5 | 91.4
  AASLD Criteria | 80.7 | 86.5
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Central Laboratory Criteria; Test type: Superiority; p = 0.2803, Cochran-Mantel-Haenszel — P-value was from CMH tests stratified by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata; Difference in the Percentages = -2.9, 95% CI 2-sided [-8.4 to 2.6] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: TAF 25 mg vs TDF 300 mg; AASLD Criteria; Test type: Superiority; p = 0.0788, Cochran-Mantel-Haenszel — P-value was from CMH tests stratified by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata; Difference in the Percentages = -5.9, 95% CI 2-sided [-12.6 to 0.7] — [estimate comment as in outcome 5, analysis 1]

18. Secondary Outcome: Percentage of Participants With Normalized ALT at Week 96 (by Central Laboratory and AASLD Criteria)
Description: as for outcome 16
Time Frame: Week 96
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 52 | 53
percentage of participants
  Central Laboratory Criteria: number analyzed (Participants) | 32 | 19
  Central Laboratory Criteria | 56.3 | 78.9
  AASLD Criteria | 55.8 | 73.6
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Central Laboratory Criteria; Test type: Superiority; p = 0.0880, Cochran-Mantel-Haenszel — P-value was from CMH tests stratified by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata; Difference in the Percentages = -23.9, 95% CI 2-sided [-51.2 to 3.4] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: TAF 25 mg vs TDF 300 mg; AASLD Criteria; Test type: Superiority; p = 0.0510, Cochran-Mantel-Haenszel — P-value was from CMH tests stratified by baseline age groups (< 50, ≥ 50 years) and baseline HBeAg status strata; Difference in the Percentages = -18.6, 95.0% CI 2-sided [-37.4 to 0.2] — [estimate comment as in outcome 5, analysis 1]

19. Secondary Outcome: Change From Baseline in FibroTest® Score at Week 48
Description: The FibroTest score is used to assess liver fibrosis. Scores range from 0.00 to 1.00, with higher scores indicating a greater degree of fibrosis. Change from baseline was calculated as the value at Week 48 minus the value at Baseline.
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed. Participants were analyzed according to the treatment to which they were randomized.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 234 | 236
scores on a scale | -0.02 (0.082) | -0.01 (0.082)
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; P-value, difference in least squares mean (LSM), and its 95% CI were derived from analysis of variance (ANOVA) model with baseline age groups (< 50, ≥ 50 years), baseline HBeAg status, and treatment group as fixed effects in the model; Test type: Superiority; p = 0.0186, ANOVA; Difference in LSM = -0.02, 95% CI 2-sided [-0.03 to 0.00]

20. Secondary Outcome: Change From Baseline in FibroTest® Score at Week 96
Description: The FibroTest score is used to assess liver fibrosis. Scores range from 0.00 to 1.00, with higher scores indicating a greater degree of fibrosis. Change from baseline was calculated as the value at Week 96 minus the value at Baseline.
Time Frame: Baseline; Week 96
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 231 | 232
scores on a scale | -0.03 (0.080) | -0.03 (0.090)
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; P-value, difference in LSM, and its 95% CI were from ANOVA with baseline age groups (<50, ≥ 50 years), baseline HBeAg status, and treatment group as fixed effects in the model; Test type: Superiority; p = 0.6956, ANOVA; Difference in LSM = 0.00, 95% CI 2-sided [-0.02 to 0.01]

21. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 48
Description: Percent Change = Change from baseline at a postbaseline visit/baseline * 100%.
Time Frame: Baseline; Week 48
Population: Participants in the Hip DXA Analysis Set (included all participants who were randomized into the study, received at least 1 dose of study drug, and had non-missing baseline hip BMD values) with available data were analysed. Participants were analyzed according to the treatment they actually received.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 225 | 226
percent change | 0.659 (2.0818) | -0.507 (1.9051)
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Difference in LSM = 1.167, 95% CI 2-sided [0.797 to 1.536]

22. Secondary Outcome: Percent Change From Baseline in Hip BMD at Week 96
Description: Percent Change = Change from baseline at a postbaseline visit/baseline * 100%.
Time Frame: Baseline; Week 96
Population: Participants in the Hip DXA Analysis Set with available data were analyzed. Participants were analyzed according to the treatment they actually received.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 227 | 224
percent change | 1.157 (2.8501) | 0.180 (2.6813)
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.0002, ANOVA; Difference in LSM = 0.977, 95% CI 2-sided [0.465 to 1.490]

23. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 48
Description: Percent Change = Change from baseline at a postbaseline visit/baseline * 100%.
Time Frame: Baseline; Week 48
Population: Participants in the Spine DXA Analysis Set (included all participants who were randomized into the study, received at least 1 dose of study drug, and had non-missing baseline spine BMD values) with available data were analysed. Participants were analyzed according to the treatment they actually received.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 227 | 229
percent change | 1.743 (3.4674) | -0.138 (3.1072)
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Difference in LSM = 1.881, 95% CI 2-sided [1.275 to 2.486]

24. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 96
Description: Percent Change = Change from baseline at a postbaseline visit/baseline * 100%.
Time Frame: Baseline; Week 96
Population: Participants in the Spine DXA Analysis Set with available data were analyzed. Participants were analyzed according to the treatment they actually received.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 229 | 227
percent change | 2.330 (3.9301) | 1.726 (3.8224)
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.0970, ANOVA; Difference in LSM = 0.604, 95% CI 2-sided [-0.110 to 1.317]

25. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate Calculated Using the Cockcroft-Gault Equation (eGFR-CG) at Week 48
Description: Cockcroft-Gault formula is as follows:
  * For men: Glomerular filtration rate (GFR) = (140 - age in years) * body weight in kg / 72 * serum creatinine (mg/dL)
  * For women: GFR = 0.85 * (140 - age in years) * body weight in kg / 72 * serum creatinine (mg/dL).
  Change from baseline was calculated as the value at Week 48 minus the value at Baseline.
Time Frame: Baseline; Week 48
Population: Participants in the Safety Analysis Set (included all randomized participants who received at least 1 dose of study drug) with available data were analyzed. Participants were analyzed according to the treatment they actually received.
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 234 | 237
mL/min | 2.240 [-3.957 to 7.704] | -1.722 [-7.020 to 2.634]
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Superiority; p < 0.0001, Wilcoxon rank sum test — P-values were from the 2-sided Wilcoxon rank sum test to compare the 2 treatment groups

26. Secondary Outcome: Change From Baseline in eGFR-CG at Week 96
Description: Cockcroft-Gault formula is as follows:
  * For men: Glomerular filtration rate (GFR) = (140 - age in years) * body weight in kg / 72 * serum creatinine (mg/dL)
  * For women: GFR = 0.85 * (140 - age in years) * body weight in kg / 72 * serum creatinine (mg/dL).
  Change from baseline was calculated as the value at Week 96 minus the value at Baseline.
Time Frame: Baseline; Week 96
Population: Participants in the Safety Analysis Set with available data were analyzed. Participants were analyzed according to the treatment they actually received.
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 232 | 232
mL/min | 1.626 [-4.580 to 6.952] | 0.544 [-5.227 to 7.678]
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; Test type: Superiority; p = 0.7535, Wilcoxon rank sum test — P-values were from the 2-sided Wilcoxon rank sum test to compare the 2 treatment groups

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: First dose date up to 161 weeks (up to approximately 3 years); Adverse Events: First dose date up to the last dose (maximum: 105 weeks) plus 3 days
Description: The Safety Analysis Set included all randomized participants who received at least 1 dose of study drug.
Groups:
- TAF 25 mg: Adverse events reported in this group occurred during the DB phase. Participants who were virologically suppressed and taking TDF 300 mg tablet orally once daily received TAF 25 mg tablet orally once daily, and placebo to match TDF once daily for up to 53 weeks in the DB phase.
- TDF 300 mg: Adverse events reported in this group occurred during the DB phase. Participants who were virologically suppressed and taking TDF 300 mg tablet orally once daily received TDF 300 mg tablet orally once daily, and placebo to match TAF once daily for up to 50 weeks in the DB phase.
- OLE TAF 25 mg From TAF 25 mg: Adverse events reported in this group occurred during the OLE phase. Participants who completed TAF treatment in the DB phase and were willing to enter in the OLE phase, received TAF 25 mg tablet orally once daily for up to 52 weeks.
- OLE TAF 25 mg From TDF 300 mg: Adverse events reported in this group occurred during the OLE phase. Participants who completed TDF treatment in the DB phase and were willing to enter in the OLE phase, received TAF 25 mg tablet orally once daily for up to 52 weeks.
Arm/Group | TAF 25 mg | TDF 300 mg | OLE TAF 25 mg From TAF 25 mg | OLE TAF 25 mg From TDF 300 mg
All-Cause Mortality (participants affected / at risk) | 0/243 | 0/245 | 0/235 | 1/237
Serious Adverse Events (participants affected / at risk) | 11/243 | 3/245 | 8/235 | 5/237
Other Adverse Events (participants affected / at risk) | 31/243 | 28/245 | 15/235 | 15/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAF 25 mg (N=243) | TDF 300 mg (N=245) | OLE TAF 25 mg From TAF 25 mg (N=235) | OLE TAF 25 mg From TDF 300 mg (N=237)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bipolar I disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Homicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAF 25 mg (N=243) | TDF 300 mg (N=245) | OLE TAF 25 mg From TAF 25 mg (N=235) | OLE TAF 25 mg From TDF 300 mg (N=237)
Upper respiratory tract infection (Infections and infestations) | 18 | 16 | 11 | 12
Nasopharyngitis (Infections and infestations) | 13 | 12 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol: Original (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT02979613/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT02979613/Prot_001.pdf
  • Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT02979613/SAP_003.pdf